CLINICAL TRIAL: NCT00146562
Title: A Phase II Study of Pegfilgrastim (Neulasta) and Darbepoetin Alfa (Aranesp) in Support of Dose-Dense Adjuvant Chemotherapy for Breast Cancer
Brief Title: Pegfilgrastim and Darbepoetin Alfa in Support of Adjuvant Chemotherapy for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harold J. Burstein, MD, PhD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Lowell General Hospital (Other); Brigham and Women's Hospital (Other); North Shore Medical Center (Other)
Responsible Party: Sponsor-Investigator, Harold J. Burstein, MD, PhD, Associate Professor of Medicine, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-154
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer
Keywords: adjuvant chemotherapy; G-CSF; pegfilgrastim; darbepoetin alfa
MeSH Terms: conditions — Breast Neoplasms | interventions — Darbepoetin alfa; pegfilgrastim; Paclitaxel; Doxorubicin; Cyclophosphamide

INTERVENTIONS:
Drug: Darbepoetin Alfa — Given day before chemotherapy of red blood cell count is below normal
  Other Names: Aranesp
Drug: Pegfilgrastim — Given as an injection the day before chemotherapy for a total of 8 injections
  Other Names: Neulasta
Drug: Paclitaxel — As part of standard adjuvant chemotherapy: Given every two weeks for 8 cycles
Drug: Doxorubicin — As part of standard adjuvant chemotherapy: Given every two weeks for 8 cycles
Drug: Cyclophosphamide — As part of standard adjuvant chemotherapy: Given every two weeks for 8 cycles

SUMMARY:
The main purpose of this study is to see if pegfilgrastim (Neulasta) is safe and useful in supporting people through dose-dense chemotherapy, and to see if a long-acting red blood cell growth factor, darbepoetin alfa(Aranesp) can reduce the need for blood transfusion in chemotherapy recipients.

DETAILED DESCRIPTION:
* Patients will receive chemotherapy every 2 weeks for up to 8 cycles (spread out of approximately 16 weeks, total) of treatment. On the day of chemotherapy treatment patients may receive an injection of darbepoetin alfa in addition to chemotherapy if their red blood cell count is below normal levels.
* On the day after chemotherapy treatment, patients will receive an injection of pegfilgrastim. There is one pegfilgrastim shot given per treatment cycle, for a total of 8 injections. Once the patient has finished chemotherapy and the last of the pegfilgrastim shots, their participation in this trial will be complete.
* While on this study the following procedures will be performed: a physical exam will be done every 2 weeks, vital signs will be done every 2 weeks, and blood tests every 2 weeks.
* This study also involves a Quality of Life Questionnaire done at the beginning of study treatment, at 2 months, 4 months, 6 months, and 1 year after starting the study treatment.
* Patients will remain on this study unless they experience unacceptable side effects from any of the treatment drugs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer clinical stage I, II or III disease. Patients must be deemed of sufficient risk for tumor or recurrence
* Patients may receive the defined adjuvant chemotherapy treatment either following definitive breast surgery or prior to definitive breast surgery
* 18 years of age or older
* ECOG performance status 0 or 1
* ANC > 1,500/uL
* Hemoglobin > 9 g/dL
* Platelets > 100,000/ul
* Total bilirubin less than or equal to ULN
* AST/ALT < 1.5 x ULN
* Creatinine within normal institutional limits
* PT/PTT < institutional upper limit of normal
* LVEF > 50%

Exclusion Criteria:

* Previous cytotoxic chemotherapy or therapeutic radiation therapy
* Pregnant or lactating women
* Receiving any other investigational agents
* Stage IV breast cancer
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pegfilgrastim or darbepoetin
* Previous exposure to G-CSF or pegfilgrastim or to recombinant erythropoetin-related growth factors.
* On antibiotics within 72 hours of registration
* Patients with immune deficiency who are at increased risk of lethal infections when treated with marrow-suppressive therapy, or HIV-positive patients receiving anti-retroviral therapy
* Sickle cell disease
* Known positive antibody response to any erythropoietic agent
* Known hematologic diseases
* Known history of hyperviscosity syndrome
* Patients on lithium
* RBC transfusion within past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2003-07; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To determine the rate of febrile neutropenia in women treated with dose-dense adjuvant chemotherapy receiving pegfilgrastim every 2 weeks. | 2 years

SECONDARY OUTCOMES:
To determine the rate of RBC transfusion among patients treated with dose-dense adjuvant chemotherapy receiving darbepoetin every 2 weeks. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Harold Burstein, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - North Shore Cancer Center, Peabody, Massachusetts